CLINICAL TRIAL: NCT04123795
Title: Multicenter, Open Label or Double-Blind, Placebo-Controlled Study to Evaluate the Pharmacokinetics, Safety, and Effectiveness of Certolizumab Pegol in Pediatric Study Participants With Moderate to Severe Chronic Plaque Psoriasis
Brief Title: A Study to Evaluate the Pharmacokinetics, Safety, and Effectiveness of Certolizumab Pegol in Children With Moderate to Severe Chronic Plaque Psoriasis
Acronym: CIMcare
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PS0007
Record Dates: First submitted 2019-10-09; First posted 2019-10-11 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Moderate Chronic Plaque Psoriasis; Severe Chronic Plaque Psoriasis; Mixed Guttate/Plaque Psoriasis
Keywords: Chronic plaque psoriasis; Certolizumab pegol; Cimzia; Pediatric study; Phase 3
MeSH Terms: interventions — Certolizumab Pegol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort A - certolizumab pegol (Experimental): Enrolling study participants aged 12 to 17 years (inclusive). Study participants in this arm will receive weight-based subcutaneous doses of certolizumab pegol from Week 1 to Week 52 of the Active Treatment period and through the subsequent Open-Label Extension Period.
  Interventions: Drug: Certolizumab pegol
- Cohort A - placebo (Placebo Comparator): Enrolling study participants aged 12 to 17 years (inclusive) under Amendment 4 and earlier. Study participants in this arm will receive weight-based subcutaneous doses of placebo from Week 1 to Week 16 of the Active Treatment period.
  Interventions: Drug: Certolizumab pegol; Drug: Placebo
- Cohort B - certolizumab pegol - Open-label (Experimental): Enrolling study participants aged 6 to 17 years (inclusive). Study participants in this arm will receive weight-based subcutaneous doses of certolizumab pegol from Week 1 to Week 52 of the Open-label Period and through the subsequent Open-Label Extension Period.
  Interventions: Drug: Certolizumab pegol

INTERVENTIONS:
Drug: Certolizumab pegol — Certolizumab Pegol
  * Pharmaceutical Form: Solution for injection in pre-filled syringe
  * Route of Administration: Subcutaneous use
  Other Names: -Cimzia; -CDP870; -CZP
Drug: Placebo — Placebo
  * Pharmaceutical Form: Solution for injection in pre-filled syringe
  * Route of Administration: Subcutaneous use
  Arms: Cohort A - placebo

SUMMARY:
The purpose of the study is to evaluate the pharmacokinetic (PK) of certolizumab pegol (CZP) in study participants aged 6 to 17 years with moderate to severe chronic plaque psoriasis (PSO) in order to support extrapolation of efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Study participant must have a diagnosis of moderate to severe plaque psoriasis (PSO) for ≥3 months and:

  1. Body Surface Area (BSA) affected by psoriasis ≥10 %
  2. Physician's Global Assessment (PGA) score ≥3 (on a scale from 0 to 4)
  3. Psoriasis Area and Severity Index (PASI) score is ≥12 or
  4. PASI score is ≥10 and <12 with at least one of the following:
* >Clinically relevant facial or scalp involvement
* >Clinically relevant genital involvement
* >Clinically relevant palm and sole involvement
* >Clinically relevant axillary involvement Study participants aged ≥12 years may alternatively have a diagnosis of moderate to severe mixed guttate/plaque PSO with >50 % to <80 % guttate lesions for ≥3 months, and must meet the same criteria listed above
* Study participant must be a candidate for systemic psoriasis therapy and/or phototherapy and/or photochemotherapy

Exclusion Criteria:

* Study participant previously participated in this study or has previously been treated with certolizumab pegol (CZP)
* Study participant has generalized pustular or erythrodermic psoriasis (PSO)
* Study participant has guttate PSO without plaque PSO
* Study participant has had a primary failure to an anti-tumor necrosis factor agent
* Study participant has had prior exposure to >2 biologic therapies
* Study participant has a history of severe major depression or suicide attempt (including an actual attempt, interrupted attempt, or aborted attempt), or has had suicidal ideation in the past 6 months as indicated by a positive response ("Yes") to either Question 4 or Question 5 of the "Screening/Baseline" version of the Columbia Suicide Severity Rating Scale (CSSRS) at Screening

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 49 (Estimated)
Dates: Start 2020-01-21 (Actual); Primary Completion 2029-09-19 (Estimated); Study Completion 2034-08-15 (Estimated)

PRIMARY OUTCOMES:
Plasma concentrations of Certolizumab pegol (CZP) at Week 16 | Week 16
  Blood samples will be collected for measurement of plasma concentrations of CZP at Week 16.
Plasma anti-CZP antibody titers at Week 16 | Week 16
  Blood samples will be collected for measurement of anti-CZP antibody titers at Week 16.
Plasma concentrations of CZP at Week 52 | Week 52
  Blood samples will be collected for measurement of plasma concentrations of CZP at Week 52.
Plasma anti-CZP antibody titers at Week 52 | Week 52
  Blood samples will be collected for measurement of anti-CZP antibody titers at Week 52.

SECONDARY OUTCOMES:
Incidence of serious treatment emergent adverse events | From Baseline until participant reaches 18 years of age or Cimzia becomes commercially available for pediatric PSO in participant's region (up to 12 years)
  A serious treatment emergent adverse event (serious TEAE) is any untoward medical occurrence that at any dose:
  * Results in death
  * Is life-threatening
  * Requires in patient hospitalization or prolongation of existing hospitalization
  * Is a congenital anomaly or birth defect
  * Is an infection that requires treatment parenteral antibiotics
  * Other important medical events which based on medical or scientific judgement may jeopardize the patients, or may require medical or surgical intervention to prevent any of the above
Incidence of treatment emergent adverse events leading to withdrawal | From Baseline until participant reaches 18 years of age or Cimzia becomes commercially available for pediatric PSO in participant's region (up to 12 years)
  An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical investigation participants administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. Treatment emergent adverse events (TEAEs) are events that emerge during treatment, having been absent pre-treatment, or worsens relative to the pre-treatment state.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (51):
- United States (41):
  - Ps0007 50214, Auburn, Alabama
  - Ps0007 50175, Phoenix, Arizona
  - Ps0007 50213, Anaheim, California
  - Ps0007 50162, Fountain Valley, California
  - Ps0007 50161, Los Angeles, California
  - Ps0007 50196, Thousand Oaks, California
  - Ps0007 50312, Aurora, Colorado
  - Ps0007 50217, Boca Raton, Florida
  - Ps0007 50248, Hialeah, Florida
  - Ps0007 50169, Jacksonville, Florida
  - Ps0007 50318, Jacksonville, Florida
  - Ps0007 50268, Miami, Florida
  - Ps0007 50216, Miami, Florida
  - Ps0007 50246, Pembroke Pines, Florida
  - Ps0007 50184, Pembroke Pines, Florida
  - Ps0007 50269, Wellington, Florida
  - Ps0007 50230, Rome, Georgia
  - Ps0007 50274, Savannah, Georgia
  - Ps0007 50168, Chicago, Illinois
  - Ps0007 50222, Overland Park, Kansas
  - Ps0007 50286, Topeka, Kansas
  - Ps0007 50188, Metairie, Louisiana
  - Ps0007 50158, Brighton, Massachusetts
  - Ps0007 50178, Clarkston, Michigan
  - Ps0007 50232, Detroit, Michigan
  - Ps0007 50186, Saint Joseph, Michigan
  - Ps0007 50105, St Louis, Missouri
  - Ps0007 50185, Lebanon, New Hampshire
  - Ps0007 50159, Newington, New Hampshire
  - Ps0007 50160, Forest Hills, New York
  - Ps0007 50247, The Bronx, New York
  - Ps0007 50229, Rocky Mount, North Carolina
  - Ps0007 50326, Marion, Ohio
  - Ps0007 50212, Tulsa, Oklahoma
  - Ps0007 50150, Philadelphia, Pennsylvania
  - Ps0007 50157, Pittsburgh, Pennsylvania
  - Ps0007 50156, Arlington, Texas
  - Ps0007 50226, Houston, Texas
  - Ps0007 50281, Laredo, Texas
  - Ps0007 50277, San Antonio, Texas
  - Ps0007 50227, Seattle, Washington
- Canada (7):
  - Ps0007 50163, Calgary
  - Ps0007 50183, Calgary
  - Ps0007 50225, Calgary
  - Ps0007 50187, Edmonton
  - Ps0007 50167, Montreal
  - Ps0007 50215, St. John's
  - Ps0007 50279, Vancouver
- Puerto Rico (3):
  - Ps0007 50231, Carolina
  - Ps0007 50278, Ponce
  - Ps0007 50265, San Juan

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: http://www.Vivli.org